CLINICAL TRIAL: NCT00964873
Title: A Phase 1 Study of the HSP90 Inhibitor, STA-9090, Administered Once-Weekly in Subjects With Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia and Blast-phase Chronic Myelogenous Leukemia
Brief Title: A Phase 1 Study of the HSP90 Inhibitor, STA-9090 in Subjects With Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia and Blast-phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-04
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Blast-phase Chronic Myelogenous Leukemia; AML; ALL; CML
Keywords: Synta; STA-9090; ganetespib; Hematologic Cancers; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Blast-phase Chronic Myelogenous Leukemia; AML; ALL; CML; HSP90 Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Part 1 (Experimental)
  Interventions: Drug: STA-9090 (ganetespib)

INTERVENTIONS:
Drug: STA-9090 (ganetespib) — Chemotherapy agent

SUMMARY:
An open-label phase 1 study to assess safety and efficacy of once-weekly STA-9090 (ganetespib) in subjects with AML, ALL and blast-phase CML.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pathologic confirmation of the diagnosis of AML, ALL, or blast-phase CML
* ECOG Performance Status 0-2
* Adequate organ function as defined in the protocol.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Hyperleukocytosis
* Acute Promyelocytic Leukemia (FAB-M3) subtype
* Uncontrolled Disseminated Intravascular Coagulation (DIC)
* Active central nervous system leukemia
* Concomitant radiation therapy, chemotherapy, or immunotherapy
* Women who are pregnant or lactating
* Neuropathy ≥ grade 2 (NCI CTCAE) at time of enrollment
* Chemotherapy (with the exception of hydroxyurea) or radiotherapy within two weeks or within six times the agent's half life
* Require ongoing therapy with either G- or GM-CSF, or long-acting versions of these molecules
* Use of any investigational agents within two weeks or within six times the agent's half life --Treatment with chronic immunosuppressants
* Other medical/psychiatric condition that may increase the risk associated with study participation as defined by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess efficacy in subjects with AML, ALL and blast-phase CML based on standard response criteria | every 8 weeks

SECONDARY OUTCOMES:
To characterize the safety and tolerability of once-weekly STA-9090 (ganetespib) in subjects with AML, ALL and blast-phase CML | ongoing
  as per adverse event and serious adverse event reporting

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Tampa, Florida
  - Baltimore, Maryland
  - Durham, North Carolina